CLINICAL TRIAL: NCT03443284
Title: A Mixed Methods Randomized, Controlled Evaluation of Health Partner mHealth for Total Joint Replacement at Providence Health & Services
Brief Title: Health Partner Evaluation at Providence
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision to close study due to low and slow enrollment.
Sponsor: DePuy Orthopaedics (Industry)
Collaborators: Johnson & Johnson Health and Wellness Solutions, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DSJ-2017-06
Record Dates: First submitted 2018-01-31; First posted 2018-02-23 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Total Knee Arthroplasty; Total Hip Arthroplasty
Keywords: Total Knee Arthroplasty; Total Hip Arthroplasty; Total Knee Replacement; Total Hip Replacement; Hospital Care Plan; mHealth
MeSH Terms: interventions — Telemedicine; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Health Partner) (Experimental): The mobile health (mHealth) product, Health Partner for Knees and Hips (Health Partner), is a combination of an iPhone or iPod Touch Operating System (iOS) mobile application (app) and a health care provider (HCP) portal.
  Interventions: Behavioral: Health Partner
- Control (Other): Patients randomized to Control will receive pre-printed brochures that outline the steps of the care plan for unilateral TKA and THA, as per standard care provided to any unilateral TJA patient receiving care at Providence Health & Services.
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Health Partner — Health Partner is a combination of an iPhone or iPod Touch Operating System mobile application and a health care provider portal.
  Other Names: mHealth
  Arms: Intervention (Health Partner)
Behavioral: Standard Care — Patients randomized to Control will receive pre-printed brochures that outline the steps of the care plan for unilateral TKA and THA, as per standard care provided to any unilateral TJA patient receiving care at Providence Health & Services.
  Other Names: Control
  Arms: Control

SUMMARY:
This is a prospective, mixed methods, multi-center, randomized, comparative, controlled study. Providence Health & Services will enroll a total of 296 subjects (18 years or older) who are electing to have total knee or hip replacement surgery. Subjects will be randomized to either the treatment group (Health Partner alongside standard care) or the control group (standard care alone). Health Partner is a combination of an iPhone or iPod Touch Operating System mobile application and a health care provider portal. The primary objective is to compare care plan adherence (pre- and post-surgery) for Health Partner vs. control subjects. Secondary objectives include evaluating all-cause medical resource utilization, communication with health care provider, well-being, fear of surgery, confidence in recovery from surgery, sleep, and patient satisfaction for 90 days post-surgery. To evaluate the behavioral factors associated with care path adherence using a qualitative interview method.To evaluate the usability and preferences of patients in their interaction with the intervention using a qualitative interview method, for product development.

The total planned study duration is approximately 1 year and 7 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 or older at the time of consent.
* Subject must be identified by their PH & S provider as needing elective unilateral TKA or THA.
* Subject is willing to give voluntary, written informed consent to participate in this Study prior to the scheduled TKA or THA surgery.
* Subject authorizes the transfer of his/her information to the Sponsor and Business Associate.
* Subject must have a valid e-mail address and willing to access their inbox on a regular basis.
* Subject must possess an iPhone/iPad/iPod Touch with operating iOS 9.0 or later and be willing to use and access digital materials from a mobile app.
* Subject must be able to comprehend and comply with the requirements of the Study.
* Subject must be able to speak, read and understand English fluently.

Exclusion Criteria:

* Subject is not able to follow the standard of care (e.g. due to allergies) and would require special care or circumstances.
* Subject scheduled to have TKA or THA sooner than 4 weeks from the time they enrolled in the study.
* Subject is undergoing a revision to a previous surgery.
* Subject is undergoing TKA or THA following traumatic injury (i.e. fracture).
* Subject is expected to need another lower limb joint replacement (hip/knee) prior to completing this Study.
* Subject is a repeat patient and was enrolled in the study previously.
* Subject has had prior experience with the Health Partner companion app.
* Subject is currently involved in any personal injury litigation, medical-legal or worker's compensation claims.
* Subject, in the opinion of the sub-investigator is a drug or alcohol abuser (in the last 5 years) or has a psychological disorder that could affect his/her ability to complete patient reported questionnaires or be compliant with follow-up requirements.
* Subject was diagnosed and is taking prescription medications to treat a muscular disorder that limits mobility due to severe stiffness and pain such as fibromyalgia or polymyalgia.
* Subject has a significant neurological or musculoskeletal disorder(s) or disease that may adversely affect gait or weight bearing activities (e.g., muscular dystrophy, multiple sclerosis, Charcot disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
Care Path Behavioral Assessment (CPBA) Pre-surgery | Early post-operative (day after surgery to 6 weeks post-surgery)
  Survey assesses degree of subject adherence with pre-surgical activities
Care Path Behavioral Assessment (CPBA), Post-surgery | Late post-operative (11-13 weeks post surgery)
  Survey assesses degree of subject adherence with post-surgical activities

SECONDARY OUTCOMES:
Medical Resource Utilization | Late post-operative (11-13 weeks post-surgery)
  Seven questions to evaluate the number and duration of encounters with the healthcare system after surgery
Confidence in Recovery (1-item) | Baseline (-6 to -3 weeks pre-surgery), pre-operative (-3 weeks to day before surgery), early post-operative (day after surgery to 6 weeks post-surgery)
  One question to guage subject's confidence in their recovery after surgery on a five-point Likert scale (ranging from Strongly disagree to Strongly sgree)
Fear of Surgery (1-item) | Baseline (-6 to -3 weeks pre-surgery), pre-operative (-3 weeks to day before surgery)
  One question to guage degree to which subject is fearful of surgery on a five-point Likert scale (ranging from Strongly disagree to Strongly sgree)
Adherence (MOS Patient Adherence) | Pre-operative (-3 weeks to day before surgery), early post-operative (day after surgery to 6 weeks post-surgery) and late post-operative (11-13 weeks post-surgery)
  The Medical Outcomes Study (MOS) Patient Adherence is a 5-item questionnaire (ranging from "None of the time" to "All of the time") guaging subject self-reported ability to follow doctors' suggestions and the frequency of subject adherence. To score general adherence, the responses are averaged together after reversing items 1 and 3.
Well-being (MQLI) | Baseline (-6 to -3 weeks pre-surgery), pre-operative (-3 weeks to day before surgery), early post-operative (day after surgery to 6 weeks post-surgery), and late post-operative (11-13 weeks post-surgery)
  The Multi-Cultural Quality of Life Index (MQLI) asks respondents to rank ten different areas of their life [self-care and independent functioning, occupational functioning, social-emotional support, community and service support, interpersonal functioning, global perception of quality of life, physical well-being, personal fulfillment, psychological/emotional well-being, and spiritual fulfillment] on a 10-point Likert scale
Well-being (PHS-WB) | Baseline (-6 to -3 weeks pre-surgery), pre-operative (-3 weeks to day before surgery), early post-operative (day after surgery to 6 weeks post-surgery), and late post-operative (11-13 weeks post-surgery)
  The Public Health Surveillance Well-Being Scale (PHS-WB) comprises 10-items guaging self-reported mental, physical, and social components of well-being. Response options for 6 of the items are on a 5-point Likert-type scale. The responses options range from "strongly disagree" to "strongly agree," "none of the time" to "all of the time," and "poor" to "excellent." Three of the items are based on a 10-point Likert-type scale. Response options for the 10-point items range from "very dissatisfied" to "very satisfied." One item assesses energy/vitality over the past 30 day. The responses for that item ranged from 0 to 30. A score for the PHS-WB scale was created by summing the 10 items for each respondent.
Sleep (MOS Sleep Scale) | Baseline (-6 to -3 weeks pre-surgery), pre-operative (-3 weeks to day before surgery), early post-operative (day after surgery to 6 weeks post-surgery), and late post-operative (11-13 weeks post-surgery)
  The MOS Sleep Scale is a 12-item instrument, which measures multiple facets of sleep. The MOS Sleep Scale yields a sleep problems index and six scale scores: sleep disturbance (have trouble falling asleep, how long to fall asleep, sleep was not quiet, awaken during your sleep time, and have trouble falling asleep again), sleep adequacy (get enough sleep to feel rested upon waking in the morning and get amount of sleep needed), daytime somnolence (drowsy during day, have trouble staying awake during the day, and take naps), snoring, awaken short of breath or with headache, and quantity of sleep. Quantity of sleep is scored as the average hours slept per night. The other scales and problems index are scored on a range from 0 to 100 with higher scores indicating more of the concept being measured.
Sleep (2-items) | Baseline (-6 to -3 weeks pre-surgery), pre-operative (-3 weeks to day before surgery), early post-operative (day after surgery to 6 weeks post-surgery), and late post-operative (11-13 weeks post-surgery)
  Two questions to assess whether subjects had 7-9 hours of restful sleep per night
Communication (1-item) | Baseline (-6 to -3 weeks pre-surgery), pre-operative (-3 weeks to day before surgery), early post-operative (day after surgery to 6 weeks post-surgery), and late post-operative (11-13 weeks post-surgery)
  One question to assess the frequency of subject's communication with their provider
Qualitative Interview | Group 1: 1-7 days pre-surgery, Group 2: 7-10 weeks post-surgery
  A qualitative interview to evaluate the behavioral factors associated with care path adherence and to evaluate the usability and preferences of patients in their interaction with the intervention, for product development.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Croy, MD, Principal Investigator — Providence Newberg Medical Center; Arnold Peterson, MD, Principal Investigator — Providence Sacred Heart/Holy Family
Locations (3):
- United States (3):
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Sacred Heart Hospital, Spokane, Washington
  - Providence Holy Family Hospital, Spokane, Washington